CLINICAL TRIAL: NCT06268782
Title: Online Training Program for Postpartum Women - How to Effectively Enhance the Well-being and Recovery After Pregnancy and Delivery
Brief Title: The Effectiveness of an Online Exercise Program on Well-being of Postpartum Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Collaborators: Finnish Cultural Foundation (Other)
Responsible Party: Principal Investigator, Iina Ryhta, Doctoral researcher, University of Turku
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1204202118
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Quality of Life; Physical Activity; Urinary Incontinence; Pelvic Organ Prolapse
Keywords: digital health intervention; ehealth; exercise; mother; physical activity; postpartum; quality of life; urinary incontinence; pelvic organ prolapse
MeSH Terms: conditions — Motor Activity; Urinary Incontinence; Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The intervention group (Experimental): All participants belonged to the intervention group. The participants were asked to answer for the pretest questionnaire before the intervention, then accomplish the six-week intervention, answer to the posttest questionnaire after the intervention and answer to the follow-up questionnaire six months after the intervention.
  Interventions: Behavioral: Rehabilitate your core

INTERVENTIONS:
Behavioral: Rehabilitate your core — The intervention was an online exercise program "Rehabilitate your core," designed for postpartum women by a company called Nordic Fit Mama. Its primary goal is to fortify the core and pelvic floor muscles to enhance the recovery process after childbirth, while also emphasizing overall well-being. The program is accessible through a website and is intended to be completed independently over a span of 6 weeks. Each week focuses on a specific theme, encompassing six to seven subtopics. The regimen follows a progressive structure, starting with the identification of pelvic floor and core muscles and gradually advancing to exercises aimed at strengthening them. The exercises, which last around 10 minutes each, are tailored to integrate seamlessly into daily life. Comprising 25 instructional exercise videos and 13 guidance videos, the program only necessitates access to a device for logging into the platform.

SUMMARY:
The aim of this quasi-experimental study was to assess the effectiveness of a 6-week online exercise program on self-assessed quality of life (QoL), physical activity (PA), and dysfunctions of pelvic floor muscles of postpartum women immediately and 6 months after the online intervention. The data were collected with e-questionnaires. The data collection started in September 2021 and ended in September 2023.

DETAILED DESCRIPTION:
The aim of this study was to assess the effectiveness of a 6-week online exercise program on self-assessed quality of life (QoL), physical activity (PA), and symptoms of urinary incontinence (UI) and pelvic organ prolapse (POP) of postpartum women immediately and 6 months after the online intervention. The hypothesis was that the online exercise program increases PA, which consequently improves QoL and decreases the symptoms of UI and POP immediately and 6 months after the intervention.

This study was a quasi-experimental study with pre- and posttest design, without a control group. It was carried out in Finland between September 2021 and September 2023. Data were collected with e-questionnaires at the baseline (pretest), immediately after the intervention (posttest), and 6 months after the intervention (6-month follow-up). Ethical approval for this study was obtained from the Ethics Committee for Human Sciences at the University of Turku in June 2021.

The intervention was a Finnish-language online exercise program "Rehabilitate your core" developed for postpartum women by a company called Nordic Fit Mama. The program aims to strengthen the core and pelvic floor muscles for enhancing recovery after pregnancy and birth, but overall well-being is also considered throughout the program. The program is built on a webpage and is planned to be accomplished independently in 6 weeks. Every week has a specific theme, which includes six to seven subthemes. The program is progressive.

The study participants were recruited via the webpage of the online exercise program and every person participating in the online exercise program between September 2021 and January 2023 were invited to participate in this study. The eligibility criteria were: an age ≥18; a maximum of 2 years from the last birth; a complete postnatal examination (usually done 5-12 weeks after birth); fluency in Finnish; and the ability to pay for access to the online exercise program.

The sample size was determined by the WHOQOL-BREF instrument used in previous studies, as QoL was the primary outcome of this study. Based on power analysis, a total of 127 participants were required to detect a difference between baseline, pretest, and posttest measures. Considering the loss to follow-up, the sample size was increased to 303 at the baseline.

Data were collected with REDCap e-questionnaires that consisted of demographic data and validated instruments (The World Health Organization Quality of Life (WHOQOL-BREF), Physical Activity Questionnaire Short Form (IPAQ-SF), Incontinence Impact Questionnaire IIQ-7 and Urogenital distress inventory UDI-6).

Descriptive statistics (means, standard deviations or medians, frequencies, and percentages) were used to summarize the demographic data. The statistical analysis of the changes of mean or median scores of primary and secondary outcomes were tested using the Wilcoxon signed-rank test or paired samples t-test. Correlations between demographic data and the outcomes were tested with Pearsons and Spearmans correlations, the independent samples t-test, the Mann-Whitney U test, the one-way ANOVA, or the Kruskal-Wallis tests. The level of statistical significance was set at p≤.05. The data were analyzed using the IBM SPSS Statistics® program, version 28.

ELIGIBILITY:
Inclusion Criteria:

* a maximum of 2 years from the last birth
* a complete postnatal examination (usually 5-12 weeks after birth)
* the ability to pay for access to the online exercise program
* fluency in Finnish

Exclusion Criteria:

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2023-01-24 (Actual); Study Completion 2023-09-19 (Actual)

PRIMARY OUTCOMES:
Quality of Life | From enrollment to the end of follow-up period 6 months after the intervention
  The primary outcome, quality of life, was measured with The World Health Organization Quality of Life (WHOQOL-BREF) instrument. The WHOQOL-BREF is a 26-item assessment instrument, which purpose is to assess individuals' perceptions of their position in life relation to their goals, expectations, standards and concerns. The first two items of WHOQOL-BREF measure the overall QoL and general health. The rest of the items of WHOQOL-BREF are divided into four different domains: physical health (7 items), psychological health (6 items), social relationships (3 items), and environment (8 items). Each item is rated on a 5-point Likert scale (a low score of 1 to a high score of 5). Data were analyzed according to the scoring guideline. During the data processing, the raw item score of each domain was calculated, and then the domain raw scores were converted to a scale from 0 to 100, where a higher score represented a higher QoL.

SECONDARY OUTCOMES:
Physical activity | From enrollment to the end of follow-up period 6 months after the intervention
  PA was measured with the International Physical Activity Questionnaire Short Form (IPAQ-SF) instrument. The IPAQ-SF is a 7-item assessment instrument whose purpose is to assess the types of the intensity of PA and sitting time that people perform as a part of their daily lives. Participants were asked to address the number of days and the time that they spent on PA in moderate and vigorous intensity and walking during the last 7 days. The scores are expressed in PA metabolic equivalent of task (MET) minutes per week. Time spent sitting is calculated as time per day and week. Data from IPAQ-SF were analyzed according to the scoring guideline so, that in the end of the data processing the data related to PA were described as followed: walking MET minutes per week, moderate MET minutes per week, vigorous MET minutes per week and total MET minutes per week.
Urinary incontinence | From enrollment to the end of follow-up period 6 months after the intervention
  The urinary incontinence was measured with two instruments that are recommended to use together: Incontinence Impact Questionnaire IIQ-7 (short version of the original instrument) and Urogenital distress inventory UDI-6 (short version of the original instrument). These two instruments include altogether 13 items with Likert scales (with item responses 0 for "not at all" to 3 "greatly") and the instruments are used to research the impact on the quality of life of incontinence symptoms in women.
Pelvic organ prolapse | From enrollment to the end of follow-up period 6 months after the intervention
  Symptoms of pelvic organ prolapse were measured with five questions. There were three questions regarding the prevalence of prolapse symptoms with options yes/no, which were retrieved from the Urogenital distress inventory -instrument's full version, and two questions evaluated with VAS, which goal were to assess the severity of the symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Axelin, PhD, Study Director — University of Turku
Locations (1):
- Department of Nursing Science, Faculty of Medicine, University of Turku, Turku, Finland

IPD SHARING:
Plan to Share IPD: No
The data that we collected were really personal and sensitive and the participants were considered as vulnerable group as study participants, so we decided not to share the data.